CLINICAL TRIAL: NCT02338037
Title: An Intracerebral Microdialysis Study to Determine the Neuropharmacokinetics of Eribulin in Patients With Brain Tumors
Brief Title: Neuropharmacokinetics of Eribulin Mesylate in Treating Patients With Primary or Metastatic Brain Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14312; NCI-2014-02391 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14312 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-12-03; First posted 2015-01-14 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Malignant Neoplasm in the Adult Brain; Primary Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Biopsy; eribulin; Microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (eribulin mesylate) (Experimental): Patients undergo tumor resection or biopsy and have microdialysis catheter placed on day 0. Beginning at least 24 hours later, patients receive eribulin mesylate IV over 2-5 minutes on day 1. Serial brain fluid samples are collected for approximately 72 hours and the microdialysis catheter is then removed. Beginning at least 2 weeks after tumor resection or biopsy, patients may continue to receive eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Therapeutic Conventional Surgery; Procedure: Biopsy; Drug: Eribulin Mesylate; Procedure: Microdialysis; Other: Pharmacological Study

INTERVENTIONS:
Procedure: Therapeutic Conventional Surgery — Undergo tumor resection
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Drug: Eribulin Mesylate — Given IV
  Other Names: E7389; ER-086526
Procedure: Microdialysis — Undergo intracerebral microdialysis
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This pilot trial studies the brain concentration of eribulin mesylate in treating patients with primary or metastatic brain tumors. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Collecting small samples of brain fluids may help determine how well eribulin mesylate concentrates into the brain tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the neuropharmacokinetic (nPK) profile of eribulin (eribulin mesylate) using intracerebral microdialysis.

SECONDARY OBJECTIVES:

I. To compare concentrations of eribulin in tumor (enhancing tissue) and normal brain (non-enhancing tissue) when technically feasible to place two microdialysis catheters in a study patient.

II. To describe the intracerebral clinical benefit (defined as stable disease, partial response, or complete response) of eribulin in study patients who continue to be treated with eribulin after completing the microdialysis portion of the study.

III. To document the toxicity of eribulin in the cohort of patients.

OUTLINE:

Patients undergo tumor resection or biopsy and have microdialysis catheter placed on day 0. Beginning at least 24 hours later, patients receive eribulin mesylate intravenously (IV) over 2-5 minutes on day 1. Serial brain fluid samples are collected for approximately 72 hours and the microdialysis catheter is then removed. Beginning at least 2 weeks after tumor resection or biopsy, patients may continue to receive eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Karnofsky performance status of >= 60
* Brain tumor patient is planning to undergo tumor resection or biopsy for the purpose of differentiating between tumor progression versus treatment-induced effects following radiation therapy and/or chemotherapy

  * If a patient has magnetic resonance imaging (MRI) findings consistent with tumor but does not already have a histopathologic diagnosis of cancer, s/he may sign the consent form, but final eligibility for study enrollment will be determined based on results of the frozen section at time of surgery
* Patient may have received previous treatment for the brain tumor(s), including radiation (focal brain radiation, whole brain radiation or stereotactic radiosurgery), surgery or chemotherapy
* There is no limit to the number of prior chemotherapies
* Patients who have previously been treated with eribulin are allowed to participate in the microdialysis portion of the study only
* Absolute neutrophil count of > 1500 cells/mm^3
* Platelet count > 100,000 cells/mm^3
* Total bilirubin < 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 3 times the institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 times the institutional upper limit of normal
* Serum creatinine < 1.5 x the institutional upper limit of normal
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients must have sufficiently recovered (=< grade 1) from any toxicity of prior therapy; the required waiting period between the last dose of the most recent chemotherapy agent and the first dose of eribulin will be determined based on the half-life of the chemotherapy agent; the minimum time between stopping prior therapy and administering the first dose of eribulin should be 3.3 half-lives with the following exceptions: an interval of at least 6 weeks must elapse since treatment with a nitrosourea and at least 4 weeks since the last dose of bevacizumab
* If corticosteroids are required for controlling cerebral edema, patients must be on a stable dose of at least 1 week prior to enrollment
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for 3 months following duration of study participation; women of child-bearing potential must have a negative serum pregnancy test prior to enrollment; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Patients who are currently receiving chemotherapy, radiation therapy or are enrolled in another therapeutic clinical trial
* Patients who have not recovered from the toxicities of prior chemotherapy or radiation
* Patients who are taking any of the prohibited medications; if a patient is willing to discontinue such a medication in order to participate in the study, then there must be an appropriate washout period, based on the half-life of the particular drug, prior to the start of the study treatment
* Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines, unstable angina or myocardial infarction within the previous 6 months
* Clinically significant cardiac arrhythmias, prolonged QT interval, congenital long QT syndrome
* Patients who cannot undergo brain magnetic resonance imaging (MRIs)
* Patients with existing grade 3 or 4 peripheral neuropathy
* Patients who have a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol or may not be able to comply with the safety monitoring requirements of the study
* Female patients who are pregnant or breast-feeding
* Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals
* Non-compliance: subjects who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-05-19 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Time of maximum concentration observed (Tmax) for eribulin mesylate | Baseline, at 5, 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48, and 72 hours and then 1 week after the infusion of eribulin mesylate
  Pharmacokinetic data will be summarized by using descriptive statistics and graphical methods. The pharmacokinetic parameters will be calculated on the log scale along with means and 95% confidence limits based on a t distribution.
Maximum concentration observed (Cmax) for eribulin mesylate | Baseline, at 5, 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48, and 72 hours and then 1 week after the infusion of eribulin mesylate
  Pharmacokinetic data will be summarized by using descriptive statistics and graphical methods. The pharmacokinetic parameters will be calculated on the log scale along with means and 95% confidence limits based on a t distribution.
Area under the curve (AUC) for eribulin mesylate | Baseline, at 5, 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48, and 72 hours and then 1 week after the infusion of eribulin mesylate
  Pharmacokinetic data will be summarized by using descriptive statistics and graphical methods. The pharmacokinetic parameters will be calculated on the log scale along with means and 95% confidence limits based on a t distribution.
Half-life (t1/2) for eribulin mesylate | Baseline, at 5, 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48, and 72 hours and then 1 week after the infusion of eribulin mesylate
Ratio of AUC of eribulin mesylate in dialysate to plasma | Baseline, at 5, 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48, and 72 hours and then 1 week after the infusion of eribulin mesylate

SECONDARY OUTCOMES:
Toxicity profile of eribulin mesylate graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days
  Will be summarized in tabular form by adverse event category, grade, and attribution.
Clinical benefit rate defined as tumor response on brain MRI results | Up to 30 days
  Clinical benefit rate and associated 95% confidence limits will be calculated based on data from participants that receive at least 2 courses of eribulin mesylate.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Eroglu Z, Synold T, Badie B, Liu A, Chowdhury A, Kilpatrick J, Blanchard S, Portnow J. An intracerebral microdialysis study to determine the neuropharmacokinetics of eribulin in patients with metastatic or primary brain tumors. Cancer Chemother Pharmacol. 2024 Dec;94(6):807-813. doi: 10.1007/s00280-024-04711-2. Epub 2024 Oct 18. PMID 39422741